CLINICAL TRIAL: NCT00854009
Title: Ascending Single Dose Study of the Safety, Tolerability, and Pharmacokinetics of BLI-489 Administered Intravenously to Healthy Japanese Male Subjects
Brief Title: Study Evaluating Single Doses of BLI-489 in Healthy Japanese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3219K1-1004
Record Dates: First submitted 2009-02-13; First posted 2009-03-02 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Healthy
Keywords: Healthy Subjects
MeSH Terms: interventions — BLI-489

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): BLI-489
  Interventions: Drug: BLI-489
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BLI-489
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single doses of BLI-489 administered intravenously in healthy Japanese male subjects, and how the drug is absorbed and eliminated.

ELIGIBILITY:
Inclusion Criteria:

1. Men, aged 20 to 50 years of age inclusive at screening.
2. Body mass index (BMI) in the range of 17.6 to 26.4 kg/m2 and body weight ≥45 kg.
3. Healthy as determined by the investigator on the basis of the screening evaluations.
4. Nonsmoker of smoker of fewer than 10 cigarettes per day as determined by history.

Exclusion Criteria:

1. Presence of history of any disorder that may prevent the successful completion of the study.
2. History of drug abuse within 1 year.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-02-20 (Actual); Primary Completion 2009-04-01 (Actual); Study Completion 2009-04-27 (Actual)

PRIMARY OUTCOMES:
Safety as measured by the number of adverse events and serious adverse events. Tolerability will be assessed based upon the occurrence of dose limiting toxicities. | 15 days

SECONDARY OUTCOMES:
Pharmacokinetics as evaluated by drug concentrations in the blood and urine. | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Tokyo, Japan